CLINICAL TRIAL: NCT05837832
Title: Phospholipids as Nutritional Support for Reduction of Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 192-002
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Participants will consume the dietary supplement every morning for 4 weeks.
  Interventions: Dietary Supplement: Milk-based phospholipids

INTERVENTIONS:
Dietary Supplement: Milk-based phospholipids — Powder based, fat-rich fraction of whey dissolved in water. Contains lactose.

SUMMARY:
The goal of this clinical trial is to learn about the effects of a milk-based dietary supplement in adults that report regular and frequent episodes of intermittent anxiety. The main question it aims to answer is: Can this extract be used to reduced symptoms of intermittent anxiety?

Participants will consume the milk-based dietary supplement every morning for 4 weeks and each week they will fill out 3 different questionnaires.

DETAILED DESCRIPTION:
Clinical study evaluating the effects of a dietary milk-based supplement to help reduce symptoms of anxiety. The milk-based supplement is a fat-rich fraction of whey, rich in phospholipids.

24 subjects who report frequent and regular episodes of intermittent anxiety will participate in a questionnaire based clinical trial, wherein they will be consuming the milk-based dietary supplement each morning for 4 weeks.

Each week subjects will fill out 2 questionnaires evaluating their anxiety and 1 questionnaire evaluating their sleep. Changes in stress will be measured relative to baseline scores, collected during the first week before supplement consumption.

ELIGIBILITY:
Inclusion Criteria:

* Adult people of any gender
* Age 18-75 years (inclusive)
* BMI between 18.0 and 34.0 (inclusive)
* Experiencing intermittent episodes of anxiety on a regular basis, leading to either avoiding specific situations, or experiencing stress both in anticipation of, and during such situations.
* Specific situations that occur regularly that cause anxiety, for example:
* Performing specific tasks at work or at home
* Inter-personal conflicts at work or at home
* Driving or commuting
* Fearful and worrying about one's own situation (such as paying bills)
* Worrying about ongoing problems experienced by others

Exclusion Criteria:

* Cancer during the past 12 months
* Chemotherapy during the past 12 months
* Currently taking anxiolytic, hypnotic, or anti-depressant prescription medication
* Currently taking nutritional supplements judged by the study coordinator to negate or camouflage the effects of the test product
* Food allergies or insensitivity related to lactose or other ingredients in test product
* People who are pregnant, nursing, or trying to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
General Anxiety Disorder-7 (GAD-7) Questionnaire | 1 week, 2 weeks, 3 weeks, 4 weeks
  Change from baseline in anxiety score using the General Anxiety Disorder 7-item. The General Anxiety Disorder-7 scale evaluates anxiety severity using scores ranging from 0-21, higher scores indicate higher anxiety severity, a worse outcome.

SECONDARY OUTCOMES:
Overall Anxiety Severity and Impairment Scale (OASIS) Questionnaire | 1 week, 2 weeks, 3 weeks, 4 weeks
  Change from baseline in Overall Anxiety Severity and Impairment Scale (OASIS) score. The Overall Anxiety Severity and Impairment scale evaluates anxiety and fear in participants with a score between 0 and 25, higher scores indicate higher anxiety severity, a worse outcome.

OTHER OUTCOMES:
Leeds Sleep Evaluation | 1 week, 2 weeks, 3 weeks, 4 weeks
  Changes from baseline in sleep quality

IPD SHARING:
Plan to Share IPD: No